CLINICAL TRIAL: NCT02589028
Title: The Effects of Premeal Consumption of Protein-enriched Bar on Blood Glucose Level and Secretion of Hormones in Healthy Adults and Patients With Type 2 Diabetes
Brief Title: The Effects of Premeal Consumption of Protein-enriched Bar on Blood Glucose Level and Secretion of Hormones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H-1504-103-666
Record Dates: First submitted 2015-10-26; First posted 2015-10-28 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2015-10

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; incretin hormone; glucose level; GLP-1; GIP; premeal protein
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- premeal protein bar first (Experimental): intervention: premeal protein-enriched bar intake
  * protein enriched bar(total serving: 30g, 43.28% carbohydrate; 1.29% fat; 40.39% protein; 42.63% fiber) will be given 30 minutes before breakfast
  * protein enriched bar is provided with 150 ml of water
  * amount of protein bar : 30g
  * breakfast : plain bagel, cream cheese, strawberry jam, orange juice 210ml
  Interventions: Dietary Supplement: premeal protein-enriched bar intake
- breakfast first (Other): intervention: breakfast follows by protein bar
  * protein enriched bar is provided with 150 ml of water shortly after breakfast
  * amount of protein bar : 30g
  * breakfast : plain bagel, cream cheese, strawberry jam, orange juice 210ml
  Interventions: Other: breakfast follows by protein bar

INTERVENTIONS:
Dietary Supplement: premeal protein-enriched bar intake — Premeal protein bar is provided 30 minutes before breakfast. Participants have to eat protein bar with in 5 minutes with 150ml of water.
  Other Names: premeal protein bar
  Arms: premeal protein bar first
Other: breakfast follows by protein bar — Participants have to eat provided breakfast within 30 minutes. It is recommended for participants to eat protein bar shortly after finishing breakfast within 5 minutes.
  Arms: breakfast first

SUMMARY:
The aim of this study is to explore premeal protein-enriched bar effect in postprandial glucose levels and concentration of plasma incretin hormones [glucagon-like peptide 1 (GLP-1) and/or glucose-dependent insulinotropic polypeptide (GIP)] in healthy subjects and those with type 2 diabetes.

DETAILED DESCRIPTION:
Fifteen healthy subjects and fifteen subjects with type 2 diabetes treated by diet and/or metformin, SU, DPP4 inhibitors will be recruited. Every subject will studied on 2 separate days in random order with 1-2 week intervals. These participants will consume protein enriched bar followed by a standardized high-glycemic-index breakfast in a hospital setting or breakfast followed protein enriched bar in a cross-over fashion. Blood sampling will be done at the moment of start of breakfast (0 min) and then 10, 20, 30, 60, 90, 120, 150, 180 min. Plasma glucose levels, total/active GLP-1, GIP, insulin, C-peptide, glucagon will be measured. Incremental area under the curve (iAUC) of glucose level and hormone from 0 min to 180 min will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5~35 kg/m2
* Healthy volunteer:

  * never diagnosed by diabetes and
  * fasting plasma glucose <=100mg/dl and HbA1c <6.0%
* participants with diabetes

  * diagnosed by diabetes
  * if treated by diet, HbA1c 6.0~9.0%
  * if treated by metformin or SU, HbA1c 6.0~10.0%
  * if treated by DPP4 inhibitor HbA1c 6.0~9.0%

Exclusion Criteria:

* Those who diagnosed by Type 1 diabetes
* History of DKA
* History of insulin therapy
* Allergy to wheat, flour, nuts, milk
* Pregnancy/lactation
* AST or ALT >2.5 times of upper normal reference range
* eGFR <30 mL/min/1.73m2
* Hb <10g/dl
* History of GI surgery (except hemorrhoidectomy, appendectomy)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
plasma glucose level after breakfast | -30 min, 0(breakfast), 10, 20, 30, 60, 90, 120, 150, 180min
Area under the curve (AUC) of plasma glucose level after breakfast | -30 min, 0(breakfast), 10, 20, 30, 60, 90, 120, 150, 180min

SECONDARY OUTCOMES:
plasma total/active GLP-1 level after breakfast | -30 min, 0(breakfast), 10, 20, 30, 60, 90, 120, 150, 180min
Area under the curve of plasma total/active GLP-1 level after breakfast | -30 min, 0(breakfast), 10, 20, 30, 60, 90, 120, 150, 180min
plasma GIP level after breakfast | -30 min, 0(breakfast), 10, 20, 30, 60, 90, 120, 150, 180min
Area under the curve of plasma GIP level after breakfast | -30 min, 0(breakfast), 10, 20, 30, 60, 90, 120, 150, 180min
plasma insulin level after breakfast | -30 min, 0(breakfast), 10, 20, 30, 60, 90, 120, 150, 180min
Area under the curve of plasma insulin level after breakfast | -30 min, 0(breakfast), 10, 20, 30, 60, 90, 120, 150, 180min
plasma C-peptide level after breakfast | -30 min, 0(breakfast), 10, 20, 30, 60, 90, 120, 150, 180min
Area under the curve of plasma C-peptide level after breakfast | -30 min, 0(breakfast), 10, 20, 30, 60, 90, 120, 150, 180min
plasma glucagon level after breakfast | -30 min, 0(breakfast), 10, 20, 30, 60, 90, 120, 150, 180min
Area under the curve of plasma glucagon level after breakfast | -30 min, 0(breakfast), 10, 20, 30, 60, 90, 120, 150, 180min

CONTACTS AND LOCATIONS:
Overall Officials: Young Min Cho, MD, PHD, Study Chair — Associate Professor Division of Endocrinology and Metabolism Department of Internal Medicine Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea